CLINICAL TRIAL: NCT06093568
Title: Exploring Engagement Dynamics Among Individuals Impacted by Renal Cell Carcinoma
Brief Title: Delving Into Participation Trends in Renal Cell Carcinoma Studies
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 74504682
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study seeks to delve into the firsthand experiences of patients diagnosed with renal cell carcinoma who partake in a separate clinical study featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

By joining this clinical trial, individuals have the unique opportunity to contribute to the betterment of future renal cell carcinoma patients and play an active role in advancing clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with renal cell carcinoma
* Patient is a minimum of 18 years or older
* Patient has self-identified as planning to enroll in a clinical study

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Inability to perform regular electronic reporting
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with renal cell carcinoma who are actively considering enrolling in an observational clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a renal cell carcinoma clinical study | 3 months
Rate of patients who remain in renal cell carcinoma clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Petejova N, Martinek A. Renal cell carcinoma: Review of etiology, pathophysiology and risk factors. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2016 Jun;160(2):183-94. doi: 10.5507/bp.2015.050. Epub 2015 Nov 3. PMID 26558360
- [Background] Bakouny Z, El Zarif T, Dudani S, Connor Wells J, Gan CL, Donskov F, Shapiro J, Davis ID, Parnis F, Ravi P, Steinharter JA, Agarwal N, Alva A, Wood L, Kapoor A, Ruiz Morales JM, Kollmannsberger C, Beuselinck B, Xie W, Heng DYC, Choueiri TK. Upfront Cytoreductive Nephrectomy for Metastatic Renal Cell Carcinoma Treated with Immune Checkpoint Inhibitors or Targeted Therapy: An Observational Study from the International Metastatic Renal Cell Carcinoma Database Consortium. Eur Urol. 2023 Feb;83(2):145-151. doi: 10.1016/j.eururo.2022.10.004. Epub 2022 Oct 20. PMID 36272943
- [Background] Schmidinger M, Bamias A, Procopio G, Hawkins R, Sanchez AR, Vazquez S, Srihari N, Kalofonos H, Bono P, Pisal CB, Hirschberg Y, Dezzani L, Ahmad Q, Jonasch E; PRINCIPAL Study Group. Prospective Observational Study of Pazopanib in Patients with Advanced Renal Cell Carcinoma (PRINCIPAL Study). Oncologist. 2019 Apr;24(4):491-497. doi: 10.1634/theoncologist.2018-0787. Epub 2019 Mar 13. PMID 30867244

DOCUMENTS (1):
  • Informed Consent Form (2023-10-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT06093568/ICF_000.pdf